CLINICAL TRIAL: NCT04368455
Title: Increasing HPV Vaccination Rates Through Virtual Immersive Communication Training on Recommending Immunizations: An Efficacy Study of VICTORI
Brief Title: Virtual Immersive Communication Training on Recommending Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brittany Rosen (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Brittany Rosen, Assistant Professor, University of Cincinnati Department of Pediatrics, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-0829; 5R21CA238170-02 (NIH)
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Human Papilloma Virus
Keywords: Human Papilloma Virus; Human Papilloma Virus Vaccine; Virtual reality; Simulation-based medical education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Care Clinic (Experimental): Physician participants will receive the self-directed app based curriculum. The physician participants will engage in the VR simulations independently.Next, we will implement VICTORI with staff including nurses and medical assistants in groups of up to 15-20 participants (phase II; secondary outcome). Staff will watch a 5-minute video on evidence-based practices in recommending the HPV vaccine and observe a facilitator and clinician participating in the VICTORI VR simulations, and then engage in a 5-minute debriefing.
  Interventions: Behavioral: Virtual Immersive Communication Training on Recommending Immunizations (VICTORI)
- Control Primary Care Clinic (Active Comparator): Physician participants will receive the self-directed app based curriculum component of VICTORI though will not undergo the VR simulations.
  Interventions: Behavioral: HPV Same Way Same Day App

INTERVENTIONS:
Behavioral: Virtual Immersive Communication Training on Recommending Immunizations (VICTORI) — An intervention that includes a self-directed app based curriculum and virtual reality simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians.
  Arms: Primary Care Clinic
Behavioral: HPV Same Way Same Day App — An intervention that includes a self-directed app based curriculum
  Arms: Control Primary Care Clinic

SUMMARY:
Our approach will be to implement Virtual Immersive Communication Training on Recommending Immunizations (VICTORI), an intervention that includes a self-directed app based curriculum and VR simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians. A single-site intervention assessing the efficacy of VICTORI in increasing HPV vaccine rates will be conducted.

DETAILED DESCRIPTION:
Background:

Despite strong evidence the human papillomavirus (HPV) vaccine is effective in preventing certain anogenital cancers, only 65% of adolescent females and 56% of males in the U.S. have initiated the series, and only 43% of girls and 31% of boys have completed it.These rates fall short of Healthy People 2020's objective of 80% coverage for adolescents years of age. Research has demonstrated that the leading predictor of parents' decisions to vaccinate their child against HPV is a strong clinician recommendation.However, evidence suggests that many parents of age-eligible adolescents are not receiving HPV vaccine recommendations or are receiving weak recommendations from clinicians.Previous interventions aimed at increasing HPV vaccination rates have had variable effects in part due to reach and adoption of the interventions within the practices. Also, the diffusion of successful interventions have been limited by lack of scalable designs.Thus, we will solve this limitation by standardizing the training component and moving towards developing a scalable model that translates into consistently improved HPV vaccine rates. Simulation-based medical education (SBME) has become an essential component of clinical training, demonstrating superior effectiveness in teaching a wide range of medical skills compared to conventional training methods. Immersive virtual reality (VR), one type of SBME, is a three-dimensional, computer-generated environment where users interact with graphical characters called avatars. Within VR, a facilitator can design scenarios based on specific behavioral objectives and create environments and avatars based on training needs. The technology facilitates deliberate practice, a personal and goal-oriented approach to skill development derived from Ericsson's Theory on Expertise. In our preliminary study conducted in 2015, we developed an intervention for resident physicians to address influenza vaccine hesitancy, comprised of a self directed application (app) based curriculum about HPV vaccination followed by immersive VR simulations.Completion of the VR simulations, compared to receipt of standard training, led to a significantly lower rate of influenza vaccine refusal.26 Based on these promising preliminary results, we developed VR simulations focused on HPV vaccine counseling.

Purpose:

Our approach will be to implement Virtual Immersive Communication Training on Recommending Immunizations (VICTORI), an intervention that includes a self-directed app based curriculum and VR simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians. VICTORI will be implemented using a framework informed by behavioral (Social Cognitive Theory, Health Belief Model, and Theory of Planned Behavior) and educational theory (Ericsson's Theory on Expertise). The primary outcome will be an increase in HPV vaccine rates among adolescent patients. We will also assess theory-based mechanisms by which the intervention changes vaccination rates, including clinicians' knowledge, attitudes, perceptions, self-efficacy, and strength of recommendations.

Our long-term goal is to increase HPV vaccination rates in adolescents, which will decrease rates of HPV-associated cancers and pre-cancers. Our short-term objective is to evaluate the efficacy of VICTORI, a novel VR intervention, designed to enhance the strength of clinicians' HPV vaccine recommendations and improve HPV vaccine rates among 11 to 17-year-old patients. To accomplish our objective, we will achieve the following specific aim:

Conduct a single-site intervention assessing the efficacy of VICTORI in increasing HPV vaccine rates. The working hypotheses are: 1) adolescent HPV vaccination rates will increase significantly following implementation of VICTORI compared to pre-intervention rates and 2) this increase will be mediated by clinicians' more positive attitudes, higher self-efficacy, and stronger vaccine recommendations.

Methods:

Clinician participants will receive a self directed app based curriculum prior to the VR simulation, VICTORI. Clinicians will receive education to increase their knowledge of HPV and the vaccine, perceived benefits, positive HPV vaccine attitudes, and subjective norms as well as decrease their perceived barriers to recommending the vaccine. The participants will engage in the VR simulations independently. VICTORI VR simulation implementation sessions will be audio and video recorded. VICTORI's effect will be assessed using a repeated measures pre-post study design with follow-up period. We will collect monthly baseline data on HPV vaccine initiation and completion rates in the clinic for six months prior to implementing VICTORI.We will then collect HPV initiation and completion rates monthly during the time of intervention implementation and for the following six-months.Next, we will implement VICTORI with staff including nurses and medical assistants in groups of up to 15-20 participants (phase II; secondary outcome). Staff will watch a 5-minute video on evidence-based practices in recommending the HPV vaccine and observe a facilitator and clinician participating in the VICTORI VR simulations, and then engage in a 5-minute debriefing. Staff will complete a brief pre and immediate post survey assessing their perceived benefits and barriers, subjective norms, and positive messaging about the HPV vaccine. We will collect an additional six months of monthly HPV vaccination initiation and completion data.

Another clinic will serve as en environmental control.Clinician participants at the control site will use the self-directed app based curriculum. Participants will complete the repeated measures pre-post study design with follow-up period. We will collect HPV vaccination data from the other primary care clinic over the same study period to serve as a control.

Implications:

The primary outcome will be the increase in the proportion of patients receiving HPV vaccination seen by resident and attending physicians following participation in VICTORI. Additional secondary outcomes, including physicians' behavioral capability, self-efficacy, perceived benefits, perceived barriers, perceived risk, attitudes, subjective norms, and strength of recommendations, as well as staffs' perceived benefits and barriers, subjective norms, and positive messaging will be assessed via validated survey instruments.

ELIGIBILITY:
Inclusion Criteria:

* Physician (Attending or Resident) at control or intervention clinic
* Staff Member (Medical Assistant or Nurse) at intervention clinic

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Joseph Real, MD, MEd, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen BL, Bishop JM, Anderson R, Real FJ, Klein MD, Kreps GL. A content analysis of HPV vaccine online continuing medical education purpose statements and learning objectives. Hum Vaccin Immunother. 2019;15(7-8):1508-1518. doi: 10.1080/21645515.2019.1587273. Epub 2019 Apr 22. PMID 30932718
- [Background] Rosen BL, Bishop JM, McDonald SL, Kahn JA, Kreps GL. Quality of Web-Based Educational Interventions for Clinicians on Human Papillomavirus Vaccine: Content and Usability Assessment. JMIR Cancer. 2018 Feb 16;4(1):e3. doi: 10.2196/cancer.9114. PMID 29453187
- [Background] Rosen BL, Shepard A, Kahn JA. US Health Care Clinicians' Knowledge, Attitudes, and Practices Regarding Human Papillomavirus Vaccination: A Qualitative Systematic Review. Acad Pediatr. 2018 Mar;18(2S):S53-S65. doi: 10.1016/j.acap.2017.10.007. PMID 29502639
- [Background] Rosen BL, Shew ML, Zimet GD, Ding L, Mullins TLK, Kahn JA. Human Papillomavirus Vaccine Sources of Information and Adolescents' Knowledge and Perceptions. Glob Pediatr Health. 2017 Nov 24;4:2333794X17743405. doi: 10.1177/2333794X17743405. eCollection 2017. PMID 29204462
- [Background] Real FJ, DeBlasio D, Ollberding NJ, Davis D, Cruse B, Mclinden D, Klein MD. Resident perspectives on communication training that utilizes immersive virtual reality. Educ Health (Abingdon). 2017 Sep-Dec;30(3):228-231. doi: 10.4103/efh.EfH_9_17. PMID 29786025
- [Background] Real FJ, DeBlasio D, Beck AF, Ollberding NJ, Davis D, Cruse B, Samaan Z, McLinden D, Klein MD. A Virtual Reality Curriculum for Pediatric Residents Decreases Rates of Influenza Vaccine Refusal. Acad Pediatr. 2017 May-Jun;17(4):431-435. doi: 10.1016/j.acap.2017.01.010. Epub 2017 Jan 23. PMID 28126612
- [Result] Real FJ, Meisman A, Rosen BL. Usability matters for virtual reality simulations teaching communication. Med Educ. 2020 Nov;54(11):1067-1068. doi: 10.1111/medu.14314. Epub 2020 Sep 10. No abstract available. PMID 32914443
- [Result] Real FJ, Ollberding NJ, Meisman AR, DeBlasio DJ, Pero MB, Davis D, Cruse B, Klein MD, Kahn JA, Rosen BL. Impact of a Virtual Reality Curriculum on Human Papillomavirus Vaccination: A Pilot Trial. Am J Prev Med. 2022 Nov;63(5):865-873. doi: 10.1016/j.amepre.2022.05.003. Epub 2022 Jun 29. PMID 35778065

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Care Clinic- Physicians: Physician participants will receive the self-directed app based curriculum. The physician participants will engage in the VR simulations independently.
  Virtual Immersive Communication Training on Recommending Immunizations (VICTORI): An intervention that includes a self-directed app based curriculum and virtual reality simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians.
- Primary Care Clinic- Staff: We will implement VICTORI with staff including nurses and medical assistants in groups of up to 15-20 participants (phase II; secondary outcome). Staff will watch a 5-minute video on evidence-based practices in recommending the HPV vaccine and observe a facilitator and clinician participating in the VICTORI VR simulations, and then engage in a 5-minute debriefing.
  Virtual Immersive Communication Training on Recommending Immunizations (VICTORI): An intervention that includes a self-directed app based curriculum and virtual reality simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians.
Period: Overall Study
Arm/Group | Primary Care Clinic- Physicians | Primary Care Clinic- Staff | Control Primary Care Clinic
Started | 97 | 27 | 37
Completed | 93 | 27 | 32
Not Completed | 4 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Analysis for providers is based upon opportunities for HPV vaccine counseling in clinic.
Groups:
- Primary Care Clinic- Physicians: Physician participants will receive the self-directed app based curriculum. The physician participants will engage in the Virtual Reality (VR) simulations independently.
  Virtual Immersive Communication Training on Recommending Immunizations (VICTORI): An intervention that includes a self-directed app based curriculum and virtual reality simulations, designed to increase the strength and consistency of human papillomavirus (HPV) vaccine recommendations among clinicians.
- Total: Total of all reporting groups
Arm/Group | Primary Care Clinic- Physicians | Primary Care Clinic- Staff | Control Primary Care Clinic | Total
Number analyzed (Participants) | 88 | 27 | 29 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing responses for age
  years
    number analyzed (Participants) | 88 | 22 | 29 | 139
    (all) | 30.1 (6.0) | 38.4 (10.8) | 32.3 (9.4) | 32.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 27 | 17 | 103
  Male | 29 | 0 | 12 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 87 | 26 | 29 | 142
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 10 | 0 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 3 | 15
  White | 66 | 16 | 20 | 102
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 5 | 1 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Percentage of Participants With HPV Vaccine Initiation
Description: The primary outcome was the percent change from pre versus post VICTORI in rates of HPV vaccine initiation among eligible patients presenting to clinic.
Time Frame: 6 months
Population: The electronic health record was used to identify patients' HPV vaccine initiation rates for participating physicians at the intervention and control sites. The pre-intervention period was 6 months before VICTORI and app-based training implementation (February 1, 2020-July 31, 2020), and the post-intervention period was 6 months following implementation (October 1, 2020-March 31, 2021). The primary outcome was the change in rates of HPV vaccine initiation pre vs post the VICTORI intervention.
Measure: Number (95% Confidence Interval); unit: Percent Change from Baseline
Groups:
- Primary Care Clinic: Physician participants will receive the self-directed app based curriculum. The physician participants will engage in the VR simulations independently entitled
  Virtual Immersive Communication Training on Recommending Immunizations (VICTORI): An intervention that includes a self-directed app based curriculum and virtual reality simulations, designed to increase the strength and consistency of HPV vaccine recommendations among clinicians.
Arm/Group | Primary Care Clinic | Control Primary Care Clinic
Number analyzed (Participants) | 88 | 29
Percent Change from Baseline | 18.1 [11.0 to 25.8] | 3.9 [-11.0 to 19.0]

2. Secondary Outcome: Physicians Perceived Barriers
Description: Physicians level barriers for recommendation of the HPV Vaccine following participation in VICTORI. Sum of 4 survey items using a 4 point scale (minimum score =4, maximum=16). A higher score indicates more barriers.
Time Frame: 3 months
Population: Secondary outcomes analyzed related to impact of curriculum over time rather than analyses compared to control participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Clinic
Number analyzed (Participants) | 75
score on a scale
  Pre-VICTORI | 7.39 (1.67)
  Post-VICTORI | 6.87 (1.66)
  3-Month Post- VICTORI | 6.75 (1.59)

3. Secondary Outcome: Physicians Perceived Risk
Description: Physicians risk of HPV for their patients following participation in VICTORI. Sum of 5 survey items using a 3 point scale (minimum score =5, maximum=15). A higher score indicates higher perceived risk for patients.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Clinic
Number analyzed (Participants) | 75
score on a scale
  Pre-VICTORI | 10.53 (2.43)
  Post-VICTORI | 12.07 (2.26)
  3 Month Post-VICTORI | 11.36 (2.36)

4. Secondary Outcome: Physicians Attitudes Toward the HPV Vaccine
Description: Physicians attitudes toward the HPV vaccine following participation in VICTORI. Sum of 12 survey items using a 5 point scale (minimum score =12, maximum=60). A higher score indicates physician perception of increased importance towards the HPV vaccine.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Clinic
Number analyzed (Participants) | 75
score on a scale
  Pre-VICTORI | 49.68 (8.73)
  Post-VICTORI | 54.24 (6.28)
  3-Month Post-VICTORI | 53.15 (7.19)

5. Secondary Outcome: Physicians Strength of Recommendation of the HPV Vaccine
Description: Physicians strength of recommendation of the HPV vaccine following participation in VICTORI. Sum of 8 survey items using a 4 point scale (minimum score =8, maximum=32). A higher score indicates stronger recommendation of HPV vaccine.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Clinic
Number analyzed (Participants) | 75
score on a scale
  Pre-VICTORI | 28.49 (3.37)
  Post-VICTORI | 28.76 (2.53)
  3-Month Post-VICTORI | 29.17 (2.35)

6. Secondary Outcome: Physicians Self-efficacy
Description: Physicians self-efficacy for recommendation of the HPV Vaccine following participation in VICTORI. Sum of 5 survey items using a 5 point scale (minimum score =2, maximum=10). A higher score indicates higher self-efficacy.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Care Clinic- Physicians
Number analyzed (Participants) | 75
score on a scale
  Pre-VICTORI | 7.44 (1.27)
  Post- VICTORI | 9.55 (0.76)
  3-Month Post-VICTORI | 9.27 (0.88)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the duration of participant participation in the research study, an average of 6 months.
Description: No adverse events occurred through study completion, an average of 6 months.
Groups:
- Primary Care Clinic- Physicians; Control Primary Care Clinic: No adverse events occurred through study completion, an average of 6 months.
- Primary Care Clinic- Staff: No adverse events occurred through study completion, one day.
Arm/Group | Primary Care Clinic- Physicians | Primary Care Clinic- Staff | Control Primary Care Clinic
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 0/88 | 0/27 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04368455/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT04368455/ICF_001.pdf